CLINICAL TRIAL: NCT01957930
Title: Intensified Insulin Treatment and Skin Microcirculation; Its Relation to Ischemic Foot Ulcer in Patients With Type 1 Diabetes Mellitus: A Long-term Follow-up Study
Brief Title: Intensive Insulin Treatment and Ischemic Foot Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Thomas Nystrom, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPI-2012
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Results first posted 2015-12-21 (Estimated); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Ischemic Foot Ulcer
Keywords: HbA1c; Iontophoresis; Intensified insulin treatment; Ischemic foot ulcer; Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intensified insulin treatment (Experimental): Basal (Monotard) insulin; ones a day Bolus (Actrapid) insulin; thrice a day
  Interventions: Drug: Intensified insulin treatment
- Standard treatment (Active Comparator): Mixed Insulin (2-3 times a day)
  Interventions: Drug: Standard treatment
- Healthy controls (No Intervention): These people were solely controls for the iontophoresis method used in the study. With no intervention or follow-up-

INTERVENTIONS:
Drug: Intensified insulin treatment — The treatment regimen of the intensified treatment group consisted of individual education and then continuous tutoring with frequent face-to-face and telephone contact.
  Other Names: Monotard; Actrapid
  Arms: Intensified insulin treatment
Drug: Standard treatment — Patients continuing with routine diabetes care (insulin treatment), visiting physician every four months
  Other Names: Premixed Insulin
  Arms: Standard treatment

SUMMARY:
We aim to investigate the relationship between skin microvascular function and the first hospitalization for ischemic foot ulcer in patients with type 1 diabetes former randomized during 7.5 years to intensified conventional insulin treatment (ICT) compared to standard insulin treatment (ST).

DETAILED DESCRIPTION:
The Stockholm Diabetes Intervention Study (SDIS) aimed to determine whether intensified insulin treatment were feasible and led to less serious diabetic complications. 102 patients with type 1 diabetes mellitus were randomiz (October 1982 to March 1984) to intensified conventional treatment (ICT; n=48) or standard treatment (ST; n=54). The randomized SDIS study lasted for 7.5 years, whereas 96 patients were fully evaluated. Thereafter patients were assigned to their regular clinical visits.

In the present study, 96 patients from the SDIS study were asked to participate in current study and to investigate their skin microcirculation, in which 72 patients agreed (ICT; n=35 vs. ST; n=37). Also, nineteen healthy subjects participated as controls for the method of iontophoresis, with no intention to be followed-up. Exclusions criteria were; any history or ongoing ischemic foot ulcer or peripheral artery disease or osteoartropathy. The iontophoresis investigation took place 5.5 years ± 2 months, after the primary randomization ceased (7.5 years). All participants (except the control subjects) were then followed-up until first time hospitalization for ischemic foot ulcer or until 31 december 2011.

ELIGIBILITY:
Inclusion Criteria:

Born 1930 or later, Type 1 diabetes appearing at age 30 or earlier and with insulin dependency within 1 year from diagnosis, no known abuse of alcohol or drugs, non-prolipherative retinopathy of any degree present, no previous photocoagulation, normal serum creatinine, unsatsifactory blood glucose control according to the physician in charge of the patients.

Exclusion Criteria:

Any history or ongoing ischemic foot ulcer,or peripheral artery disease,or osteoartropathy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 1984-01; Primary Completion 2011-12 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Nyström, MD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Karolinska Institutet, Department of Clinical Science and Education, Södersjukhuset, Stockholm
  - Karolinska Institutet, Division of Internal Medicine Södersjukhuset AB, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reichard P, Britz A, Cars I, Nilsson BY, Sobocinsky-Olsson B, Rosenqvist U. The Stockholm Diabetes Intervention Study (SDIS): 18 months' results. Acta Med Scand. 1988;224(2):115-22. doi: 10.1111/j.0954-6820.1988.tb16748.x. PMID 3048052
- [Background] Reichard P, Nilsson BY, Rosenqvist U. The effect of long-term intensified insulin treatment on the development of microvascular complications of diabetes mellitus. N Engl J Med. 1993 Jul 29;329(5):304-9. doi: 10.1056/NEJM199307293290502. PMID 8147960
- [Derived] Rathsman B, Jensen-Urstad K, Nystrom T. Intensified insulin treatment is associated with improvement in skin microcirculation and ischaemic foot ulcer in patients with type 1 diabetes mellitus: a long-term follow-up study. Diabetologia. 2014 Aug;57(8):1703-10. doi: 10.1007/s00125-014-3248-2. Epub 2014 May 7. PMID 24802206

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensified Insulin Treatment: Intensified conventional insulin treatment: The treatment regimen of the intensified treatment group consisted of individual education and then continuous tutoring with frequent face-to-face and telephone contact.
- Standard-treatment: Continuing with routine diabetes care
  Standard treatment: Patients continuing with routine diabetes care (insulin treatment), visiting physician every four months
- Healthy Controls: 19 healthy controls were invited to compare microcirculation between healthy and diabetes individuals
Period: Overall Study
Arm/Group | Intensified Insulin Treatment | Standard-treatment | Healthy Controls
Started | 35 | 37 | 19
Completed | 35 | 37 | 19
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Control: Solely controls for the iontophoresis method and no intention to be followd-up.
- Total: Total of all reporting groups
Arm/Group | Intensified Insulin Treatment | Standard-treatment | Healthy Control | Total
Number analyzed (Participants) | 35 | 37 | 19 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 35 | 37 | 19 | 91
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 42 [28 to 63] | 42 [31 to 63] | 38 [26 to 58] | 42 [28 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 8 | 51
  Male | 14 | 15 | 11 | 40
Region of Enrollment [Number; unit: participants]
  Sweden | 35 | 37 | 19 | 72

OUTCOME MEASURES:

1. Primary Outcome: Ischemic Foot Ulcer
Description: The study outcome is the first hospitalization for ischemic foot ulcer, defined by the ICD-10 discharge code
Time Frame: Until hospitalization for ischemic foot ulcer or until 31 December 2011
Population: Data for Healthy Controls was not collected for this Outcome Measure.
Measure: Number; unit: participants
Arm/Group | Intensified Insulin Treatment | Standard-treatment
Number analyzed (Participants) | 35 | 37
participants | 3 | 10

2. Other Pre Specified Outcome: Microvascular Endothelial Function
Description: Microvascular function is measured with a single point iontophoresis after stimulation with topically applied acetylcholine (ACh) [endothelial-dependent], sodium nitroprusside (SNP) [endothelial-independent], and capsaicin [C-nociceptive dependent] vasculature response.
Time Frame: 7 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Healthy Controls: These people were solely controls for the iontophoresis method used in the study. With no intervention or follow-up.
Arm/Group | Intensified Insulin Treatment | Standard-treatment | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/37 | 0/19
Other Adverse Events (participants affected / at risk) | 0/35 | 0/37 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensified Insulin Treatment (N=35) | Standard-treatment (N=37) | Healthy Controls (N=19)
0 (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes